CLINICAL TRIAL: NCT03356288
Title: An Observational Proof-of-concept Study to Explore the Waveform Characteristics of Tidal Breathing Carbon Dioxide (CO2), Measured Using the N-Tidal C™ Device, in Different Breathing Conditions.
Brief Title: The General Breathing Record Study
Acronym: GBRS
Status: Completed | Type: Observational
Sponsor: TidalSense (Industry)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: G002-17_GBRS
Record Dates: First submitted 2017-09-07; First posted 2017-11-29 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Asthma; Heart Failure; Pneumonia; Motor Neuron Disease; Vocal Cord Dysfunction; Breathlessness
Keywords: Capnography, Diagnosis. Breathlessness, Exacerbations, Device
MeSH Terms: conditions — Asthma; Heart Failure; Pneumonia; Motor Neuron Disease; Vocal Cord Dysfunction; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Asthma: 20 Participants with moderate to severe asthma, as defined by British Thoracic Society (BTS) guidelines
- Chronic heart failure: 10 Participants with a diagnosis of chronic heart failure
- Breathing Pattern Disorder: 10 Participants with a diagnosis of Breathing Pattern Disorder
- Pneumonia: 10 participants with a radiologically confirmed diagnosis of pneumonia
- Motor Neurone Disease: 10 participants with a diagnosis of motor neurone disease with known hypercapnic failure.
- Healthy: 10 Participants who have no known lung, cardiac or neuromuscular condition.

SUMMARY:
This study will test the use of a new handheld device (called the N-Tidal C), that measures a person's tidal breath carbon dioxide, in diagnosing the cause of someone's breathlessness. It will also evaluate whether this device can detect when a person's breathing problem is getting worse.

DETAILED DESCRIPTION:
When a person breathes out, they exhale carbon dioxide (CO2). The CO2 levels in breath change as they breathe out and this makes a specific pattern, or "waveform". This waveform can tell a clinician a lot about the underlying health of a person. There are disease specific CO2 waveforms for common breathing conditions such as Asthma and Chronic Obstructive Pulmonary Disease (COPD). However up until this point there has been no accurate and non-invasive method of measuring the tidal breath CO2 waveform.

This study will test the N-Tidal C, a new handheld device that accurately measures this waveform, and whether it can differentiate different causes of breathlessness; namely asthma, heart failure, pneumonia, breathing pattern disorders and motor neurone disease.

ELIGIBILITY:
Inclusion Criteria:

Asthma Cohort:

* A confirmed clinical diagnosis of asthma for ≥ 6months
* Moderate to severe asthma defined as British Thoracic Society stages 3-5
* 2 or more exacerbations in the previous 12 months with at least 1 exacerbation within the last 6 months.
* Exacerbation free for 2 weeks (defined as no increased dose or course of oral corticosteroids or antibiotics).

Breathing Pattern Disorder Cohort

* A Clinical diagnosis of a Breathing Pattern Disorder (BPD)

Chronic heart failure Cohort:

* A confirmed clinical diagnosis of chronic heart failure with both of the following:

  1. A Left Ventricular Ejection Fraction <40% on most recent imaging within the last 12 months.
  2. New York Heart Association Class 2-4
* Admitted with an acute decompensation of their heart failure to hospital within the last 6 months

Motor Neurone Disease Cohort:

* A confirmed clinical diagnosis of Motor Neurone Disease
* Forced Vital Capacity (FVC) of less than 60% of predicted, sleep disordered breathing or daytime hypercapnia.
* Established on Home Non-Invasive Ventilation.

Pneumonia Cohort:

* A confirmed clinical diagnosis of Pneumonia supported by evidence of consolidation on a chest X-ray (CXR) or computed tomography (CT) imaging.

Healthy Cohort:

* No known history of lung, cardiac or neuromuscular disease (defined as no current clinical diagnosis of, or be receiving treatment for, a lung, cardiac or neuromuscular disease). A Body Mass Index of less than 40. A Non-smoker, or an ex-smoker with less than a 5 pack year history.

Exclusion Criteria:

* Known other lung, chest wall, neuromuscular, cardiac or other comorbidity or abnormality that would affect spirometry and/or other measures of lung function or Tidal Breath Carbon Dioxide measurements.
* In the opinion of the clinical investigator, the participant would have difficulty completing the study procedures consistently over the course of 6 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The healthy Cohort will be made up of healthy volunteers. The Disease Cohorts will be selected from hospital outpatient clinic lists and inpatient wards.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
The tidal breathing carbon dioxide waveform for each of the breathing conditions as measured by the N-Tidal C device | 12 months

SECONDARY OUTCOMES:
Change in the Tidal Breathing carbon dioxide waveform over time | Change measures - baseline to 6 months
  Change in the tidal breathing carbon dioxide waveform, in each disease, over the 6 months.
Disease Control in asthma patients | 12 months
  The Asthma Control Questionnaire Score for the Asthma patients
Disease Improvement in Breathing Pattern Disorder patients | 12 months
  The Nijmegen Questionnaire Score
Disease severity in the pneumonia patients | 2 days
  The CURB-65 Score
Disease severity in heart failure patients | 12 months
  The Trans Thoracic Echocardiogram (TTE) result
Hypercapnia in the motor neurone disease patients | 12 months
  The level of partial pressure carbon dioxide (pCO2)
Usability of the N-Tidal C device | Change measures - baseline to 6 months
  Measured by how frequently the patients remember to use the N-Tidal C device over 6 months
Acceptability of the N-Tidal C device | 12 months
  Measured by a questionnaire of the participants experience of the device at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Anoop J Chauhan, PhD, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Derived] Talker L, Neville D, Wiffen L, Selim AB, Haines M, Carter JC, Broomfield H, Lim RH, Lambert G; BRS Study Team; Weiss ST, Hayward G, Brown T, Chauhan A, Patel AX. Machine diagnosis of chronic obstructive pulmonary disease using a novel fast-response capnometer. Respir Res. 2023 Jun 2;24(1):150. doi: 10.1186/s12931-023-02460-z. PMID 37268935